CLINICAL TRIAL: NCT00635713
Title: A Double-Blind, Randomized, Multi-Center Trial Comparing the Efficacy and Tolerability of 125 and 250mg of Faslodex (Long Acting ICI 182,780) With 1mg Arimidex (Anastrazole) in Postmenopausal Women With Advanced Breast Cancer.
Brief Title: Second Line Breast Cancer Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9238IL/0021; D6995C00021
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced breast cancer, FASLODEX, ARIMIDEX, Fulvestrant, Anastrozole, postmenopausal
MeSH Terms: interventions — Fulvestrant; Anastrozole

ARMS (2):
- 1 (Experimental): Faslodex 125mg and Arimidex 1 mg
  Interventions: Drug: Fulvestrant; Drug: Anastrozole
- 2 (Experimental): Faslodex 250mg and Arimidex 1mg
  Interventions: Drug: Anastrozole; Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 125mg
  Other Names: Faslodex
  Arms: 1
Drug: Anastrozole — ARIMIDEX
Drug: Fulvestrant — 250mg
  Other Names: Faslodex
  Arms: 2

SUMMARY:
The main purpose of this study is to compare the effect of 2 doses of FASLODEX with 1 dose of ARIMIDEX in terms of time to tumor progression in postmenopausal women with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with confirmation of breast cancer
* objective evidence of recurrence or progression of breast cancer no more than 1 prior hormonal therapy for breast cancer

Exclusion Criteria:

* presence of life-threatening metastatic visceral disease
* previous treatment with FASLODEX, ARIMIDEX or any aromatase inhibitor for breast cancer
* more than 1 prior endocrine medical treatment for advanced breast cancer .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 1997-05; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
time to tumor progression | Every 3 months

SECONDARY OUTCOMES:
objective tumor response | Every 3 months
time to treatment failure | Every 3 months
time to death | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Hoctin-Boes, Study Director — AstraZeneca